CLINICAL TRIAL: NCT05399862
Title: The Effect of Lactobacillus Reuteri Probiotic as an Adjunct Treatment for Helicobacter Pylori Infection in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Collaborators: Y.S.P. Industries (M) Sdn. Bhd, Menara LGB, Taman Tun Dr Ismail, 60000 Kuala Lumpur, Malaysia (Unknown)
Responsible Party: Principal Investigator, Nur Izreena Ismail, Dr, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FF-2021-004
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori, probiotics, Lactobacillus reuteri, Gastrointestinal Symptom Rating Scale, GSRS.

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients will be given Lactobacillus reuteri probiotic in addition to standard triple therapy. The probiotic is prepared in a capsule form (200mg each capsule), given as 1 capsule per day after meal for 4 weeks.
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17648 probiotic
- Group B (Placebo Comparator): Placebo used in the study contains corn starch with 0.12% of iron oxide yellow, prepared in indistinguishable capsule form as probiotic,; given as 1 capsule per day after meal for 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17648 probiotic — Lactobacillus reuteri DSM 17648 is a single-strain probiotic used as adjunct treatment in H.pylori infection
  Arms: Group A
Other: Placebo — Placebo capsule with no microbial cell preparation
  Arms: Group B

SUMMARY:
This is a prospective, randomised, double-blind, placebo-controlled trial involving newly diagnosed Helicobacter pylori (H. pylori) patients. Patients will be prescribed with standard triple therapy for 2 weeks and supplemented with either probiotic (Lactobacillus reuteri DSM 17648) or placebo for 4 weeks. In this study, we are investigating the effect of Lactobacillus reuteri in H. pylori eradication; mainly in improving eradication rate, ameliorating gastrointestinal symptoms and reducing adverse effects of antibiotics. We hypothesised that in H. pylori patients receiving Lactobacillus reuteri as adjunct treatment, there will be an improvement in H. pylori eradication rate as well as reduction of gastrointestinal symptoms and treatment adverse effects.

DETAILED DESCRIPTION:
The prime discovery of Helicobacter pylori (H. pylori) in chronic gastritis patients by Marshall and Warren in 1982 has geared a frenetic pace in H. pylori research. H. pylori is a helix-shaped microaerophilic gram negative bacterium colonising gastric epithelium leading to disruption of protective mucosal layer by inflammatory process and gastric acid secretion.

H. pylori remains as one of the commonest bacterial pathogens causing chronic infection in the adult population with at least 50% of the global population being infected. The prevalence is even higher in developing countries with up to 80% of them being affected. Although some of the patients with H. pylori infection are asymptomatic, 10-20% of them may progress into H. pylori associated disease such as chronic gastritis, peptic ulcer disease and gastric malignancy. The clinical heterogeneity is believed to be due to different degree of virulence across different H. pylori strains.

The American College of Gastroenterology (ACG) has outlined the standard therapies of H. pylori infection, dividing them into first line and salvage therapy. Treatment regime is chosen based on previous antibiotics exposure, antibiotics allergy and resistance.[7] The eradication rate of 90% is regarded as successful in which, Kyoto Global Consensus Report recommended the similar value as a cut-off point to guide the selection of empirical treatment in each region. Clarithromycin triple therapy (clarithromycin, amoxicillin/metronidazole and proton pump inhibitor, PPI) or referred as standard triple therapy (STT) in our study is recommended as first line therapy for patients who are macrolide-naive and/or reside in low clarithromycin-resistance area. For regions with high clarithromycin resistance rate (more than 15%), ACG guideline recommends administration of bismuth quadruple, non-bismuth quadruple or concomitant therapies.

The Maastricht V/Florence Consensus report has outlined the guidelines on diagnosis and therapeutic strategies in H. pylori infection. The report highlighted failure of many countries to hit at least 80% intention-to-treat eradication rate.[9] Amongst the contributing factors are emerging antibiotics resistance, poor compliance, adverse effects of antimicrobial regime leading to poor treatment adherence, high bacterial load and impairment of gastric mucosal immunity.

Regionally, the Bangkok Consensus Report by Vilaichone et al in 2018 has studied the prevalence of H. pylori infection in nine ASEAN countries. The study demonstrated high prevalence of H. pylori in ASEAN countries ranging between 20% to 69%. Despite Malaysia having the lowest H. pylori prevalence of 20%, the eradication rates failed to meet the minimum 80% target when given STT for 7 days. Qua et al (2010) and Leow et al (2018) reported the eradication rate of 71.2% and 79.3% respectively. Extending duration of STT from seven to fourteen days illustrated marked improvement of eradication rate to 88.6% but it was still below the successful eradication target of 90%.

In Malaysia, the rising primary resistance rate of H. pylori to antimicrobial agents mainly clarithromycin poses a big challenge in treating this infection effectively. The earlier studies by Teh at al (2014) demonstrated a primary resistance rate of 6.8% to both clarithromycin and fluoroquinolones, 32.3% to metronidazole; Hanafiah et al (2019) reported a primary resistance rate of 12.2%, 17.1% and 56.1% to clarithromycin, levofloxacin and metronidazole respectively. The recent study by Puah et al (2021) illustrated a further increment of clarithromycin resistance rate to 14.8%; whereas levofloxacin resistance rate was 3.3%.

Looking at the increasing antibiotics resistance and suboptimal eradication rate in Malaysia, further research to improve the overall efficacy of H. pylori eradication is undoubtedly paramount. Over the years, probiotics have shown promising benefits in a vast spectrum of gastrointestinal disorders including H. pylori infection. Several meta-analyses have demonstrated significant reduction of H. pylori eradication rate in subjects receiving probiotics as adjunct treatment. However, not all strains of probiotics are beneficial in treating H. pylori as some of them are unable to survive in the gastric environment. The Maastricht V/Florence Consensus Report emphasised that only certain probiotics are helpful in H. pylori eradication, and that includes Lactobacillus, Bifidobacterium and Saccharomyces boulardii. Amongst these, a single-strain Lactobacillus reuteri DSM 17648 has demonstrated good outcome in improving eradication rate as well as ameliorating adverse effect of treatment regime; both in human and in-vitro studies.

The probiotic used in the study was Pylobalance® which contains patented ingredient of Lactobacillus reuteri DSM 17648. The co-aggregation of probiotic and H. pylori impairs adhesion of bacterial pathogen to gastric mucosa and subsequently clears H. pylori from the stomach. The ability of Lactobacillus reuteri to co-aggregate with H. pylori without interfering with the original commensal microflora helps to preserve a stable gastric microecology. This characteristic helps to reduce gastrointestinal symptoms associated with H. pylori pathogen. The probiotic also has antimicrobial properties derived from short-chain fatty acid from lactic acid, hydrogen peroxide and bactericidal substance of reuterin which directly inhibit survival and proliferation of H. pylori. Regulation of immune response, improvement of gut mucosal barrier and production of cell-surface protein to competitively inhibit binding of H. pylori are amongst several other mechanism being proposed by previous studies to ameliorate H. pylori pathogen effect. Another advantageous characteristic of Lactobacillus reuteri is its ability to withstand unfavourable gastric environment owing to its non-viable preparation form.

To our knowledge, the efficacy of Lactobacillus reuteri probiotic as the adjunct treatment in H. pylori management has yet to be studied in Malaysian and South East Asian cohort. Owing to the clinical heterogeneity of H. pylori strains across different or even in similar population, the efficacy of Lactobacillus reuteri in our population needed to be investigated further. In this study, we sought to determine the effect of Lactobacillus reuteri in H. pylori eradication; mainly in improving eradication rate, ameliorating gastrointestinal symptoms and reducing adverse effects of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-year-old and above
* Confirmed H. pylori diagnosis
* Informed consent to participate in the study

Exclusion Criteria:

* Any active gastrointestinal disease
* Previous surgical procedures affecting the gastrointestinal tract, e.g., bariatric surgery or gastrectomy
* Pregnancy or breastfeeding women
* Previous allergy to probiotics
* Intake of proton pump inhibitor, H2 antagonist or antibiotics in the past 3 months
* Recent diagnosis of advanced stage of malignancy
* Recent acute gastroenteritis within 4 weeks
* Recent history of traditional medication intake
* Recent failure of first line eradication therapy for H. pylori

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
The eradication rate of Helicobacter pylori infection | Urea breath test is assessed at 8 weeks post treatment
  Eradication rate of H. pylori is defined as negative urea breath test result (score of less than 50 DPM)

SECONDARY OUTCOMES:
The improvement of H. pylori associated gastrointestinal symptoms | GSRS scores of both arms were compared between pre and 8 weeks post treatment
  Patient's symptoms were evaluated using Gastrointestinal Symptom Rating Scale (GSRS) which consisted of five different domains including abdominal pain, reflux, indigestion, constipation and diarrhoea
The improvement of treatment adverse effect | The treatment adverse effects were evaluated during first and second week of treatement; and further re-evaluated back at 8 weeks post treatment
  Patients were interviewed for any new adverse effects after starting the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Malaysia Medical Centre, Cheras, Kuala Lumpur, Malaysia